CLINICAL TRIAL: NCT06317519
Title: Verify the Performance in Clinical Practice of the Immersive Virtual Reality Platform GRAIL (Gait Real-time Analysis Interactive Lab) in Children and Adolescents Affected by Congenital and Acquired Brain Injury and Determine Any Secondary Effects.
Brief Title: Verify the Performance in Clinical Practice of the Immersive Virtual Reality Platform GRAIL (Gait Real-time Analysis Interactive Lab)
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2020-Oss
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Acquired Brain Injury; Cerebral Palsy
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physical Rehabilitation + GRAIL: Patients in this group receive Physical Rehabilitation and GRAIL treatment
  Interventions: Procedure: Physical Rehabilitation; Device: Gait Real-time Analysis Interactive Lab
- Physical Rehabilitation: Patients in this group receive Physical Rehabilitation not GRAIL treatment
  Interventions: Procedure: Physical Rehabilitation

INTERVENTIONS:
Procedure: Physical Rehabilitation — 5 sessions of physical rehabilitation per week. Each session lasting 45 minutes. Overall 20 sessions = 4 weeks.
Device: Gait Real-time Analysis Interactive Lab — 5 sessions of GRAIL assisted rehabilitation per week. Each session lasting 45 minutes. Overall 20 sessions = 4 weeks.
  Groups: Physical Rehabilitation + GRAIL

SUMMARY:
Gait pattern difficulties, balance and coordination deficits often characterize patients with congenital and acquired neuromotor disorders and have a significant impact on the quality of life of these subjects. There are various treatments used and in recent years, the advent of advanced technologies in rehabilitation and, in particular, devices based on virtual reality, has opened up new possibilities in rehabilitation. Virtual reality is a promising strategy that incorporates many principles crucial to motor learning, such as high-intensity, repetitive, goal-oriented tasks, enhanced synchronized sensory signals, and active participation. The virtual environment is also suitable for personalized treatment based on the needs of the individual patient.

The GRAIL (Gait Real-time Analysis Interactive Lab) is a device that integrates immersive virtual reality with an instrumented treadmill and a motion capture system, which can be used with both rehabilitation and evaluation goals. To date, there are still few studies of this device in the pediatric field.

The objective of the study is to verify the performance in clinical practice of the immersive virtual reality platform GRAIL and determine any secondary effects by evaluating whether they entail acceptable risks compared to the expected performances following the protocol defined at the IRCCS Medea by Bosisio Parini, in children and adolescents with congenital and acquired neuromotor pathology.

Patients suffering from acquired and congenital brain injuries undergo a combined rehabilitation treatment consisting of 20 sessions with GRAIL and 20 physiotherapy sessions in four weeks. The same subjects undergo evaluations before and at the end of the treatment

The study is prospective and involves the verification of performance through clinical and instrumental evaluations in the population of subjects treated with the GRAIL device at the IRCCS Medea-Bosisio Parini.

ELIGIBILITY:
Inclusion Criteria:

* Capable of following verbal requests
* Gross Motor Function Classification System score I to III

Exclusion Criteria:

* Severe spasticity
* Severe cognitive disability
* Severe auditory or visual disability

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 5 to 20 with either cerebral palsy or acquied brain injury, who can follow verbal orders and are not disabled regarding senses or intellect
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-12 (Estimated)

PRIMARY OUTCOMES:
6 minute walking test | Before and after 4 weeks of treatment
  Distance walked over 6 minutes, in meters
Gross Motor Function Measure -total score | Before and after 4 weeks of treatment
  Total score on the Gross Motor Function Measure. Greater scores indicate better performance

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS Eugenio Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No